A PROSPECTIVE RANDOMIZED STUDY COMPARING THE TIME TO HEMOSTASIS (TTH) AND SAFETY OF USING A HEMOSTASIS BAND ALONE AND IN CONJUNCTION WITH A POTASSIUM FERRATE PAD (STATSEAL ADVANCED) FOLLOWING TRANSRADIAL CATHETERIZATION.

## **Principal Investigator:**

Arnold Seto, MD, MPA
Cardiology Division
Veterans Medical Center Long Beach

NCT04046952

Original Document Date 4/2/2019

### **Table of Contents**

- I. INTRODUCTION, BACKGROUND & RATIONALE
- II. DESCRIPTION OF STUDY DEVICE
- III. STUDY OBJECTIVES
- IV. STUDY DESIGN AND METHODOLOGY
- V. STUDY ACTIVITIES AND GUIDELINES
- VI. STUDY STATISTICAL PLAN
- VII. ADVERSE EVENTS
- VIII. DATA MANAGEMENT
- IX. ETHICAL, REGULATORY AND ADMINISTRATIVE REQUIREMENTS
- X. RISK BENEFIT ANALYSIS
- XI. REFERENCES

#### **APPENDICES**

### I. INTRODUCTION, BACKGROUND & RATIONALE

Transradial access (TRA) for invasive cardiac catheterization procedures has gained significant popularity around the world compared with the transfemoral access. The 2015 European Society of Cardiology guidelines have given transradial access its highest recommendation (Class I A) over femoral access.¹ The most compelling reason for adopting TRA is the increased patient safety that results from the potential elimination of access site bleeding and vascular complications. In addition, TRA is associated with early sheath removal, improved patient comfort, faster recovery, and lower costs in comparison with transfemoral access.²-⁴ TRA provides the ability to perform a broad range of diagnostic and interventional cardiovascular procedures. In the USA, TRA catheterization procedures are gaining significant momentum with a significant growth from 2% in 507 to approximately 15% in 2011⁵, and an estimated 30- 35% in 2015. Moreover, with increased availability of training opportunities the TRA utilization rate is expected to grow to 50% or more in the next 2 – 4 years.

One important advantage of TRA is that the vascular sheath is always removed at the end of procedure regardless of the intensity of anticoagulation or antiplatelet therapy. Multiple methods for radial hemostasis have been described<sup>6</sup>. Prolonged manual compression with one or two fingers at the arteriotomy site is an effective method. Alternatively, a rolled piece of gauze can be placed longitudinally at the arteriotomy site and wrapped with an elastic bandage. These low tech, highly variable methods have been mostly abandoned in most countries in favor of inexpensive mechanical devices that apply compressive pressure to the arteriotomy site via a balloon mounted on a wrist band. These 'Hemostasis Bands' are inflated with air and apply prolonged hemostatic pressure. The disadvantage of these methods is the complete interruption of arterial flow because of the inability to gauge the hemostatic pressure applied, regardless of the methodology developed for their use. It has been demonstrated that when occlusive pressure is maintained for a period longer than two hours radial artery occlusion (RAO) occurs more often.<sup>7,8</sup> In fact, RAO after TRA procedures is not uncommon and occurs in approximately 5-10% of cases, and is accurately described as a function of time and pressure.

# Incidence RAO = ∱ (Time, Pressure)

In order to minimize the occurrence of RAO, Pancholy introduced the "patent" non-occlusive hemostasis technique, designed to address the pressure side of the RAO equation<sup>8</sup>. With this technique, a Hemostasis band is placed and a pulse oximeter is attached to the ipsilateral thumb. Then, while the sheath is being removed, the balloon is fully inflated with approximately 15-18 cc of air to completely occlude the radial artery. Subsequently, the device is slowly deflated while occlusive manual pressure is applied to the ulnar artery located at the Guyon's canal, lateral to the pisiform bone. Patent hemostasis is achieved when oximetry becomes positive and a plethysmographic waveform can be visualized. This technique assures the presence of antegrade flow in the radial artery during hemostasis. Later in recovery, small amounts of air can be periodically released, until the device is completely deflated and then removed. Using this technique, late occlusion rates can be reduced to approximately less than 5%.<sup>8</sup>

#### THE CLINICAL NEED

However, despite Pancholy's technique, meticulous patent hemostasis with careful ascertainment of adequacy of the antegrade radial flow to the hand is performed in less than

50% of cases and about a third of transradial operators are unaware of the RAO rates in their own practices.<sup>9</sup> Even when those methods<sup>10</sup>, which are recognized as being labor intensive, result in an appropriate pressure being applied, hemostasis bands are typically left in place for 2-4 hours or more in patients having undergone PCI, due to the effects of anticoagulation and the risk therein of hematoma at the access site. Because this method is labor intensive, many busy PCI programs forego this methodology in favor of alternatives, using palpable pulse methods or arbitrary inflation formulas in an attempt to achieve patent flow. In addition, the management of the band often requires actions of nursing personnel at locations outside the catheterization lab, resulting in an increased risk for complications from diminished expertise of those personnel as compared to the cath lab staff. And, even when all goes well, the impact on patient throughput and productivity when up to 4 hours of post procedure monitoring is required solely due to hemostasis band management is significant, resulting in delayed or postponed procedures, delayed discharges, additional staff expense, and other care related costs.

One method to address these deficiencies reduce the time of hemostatic compression. If radial artery compression time can be shortened to 60 minutes or less, the following could result: improved catheterization lab efficiency, greater patient satisfaction and lower complication rates, including RAO, may be improved. A system that standardizes compression technique and shortens compression time to that which is fully under the supervision and care of cath lab holding room personnel, will also eliminate the variability of recovery staff needing to manage the hemostasis band / site, and complications typically associated with patient management being carried out in multiple settings within the hospital. To summarize, the potential advantages of a hemostasis system for PCI incorporating the benefits of the StatSeal technology used in combination with a hemostasis band as compared to a hemostasis band alone may include:

- Decreased radial artery compression times, aka Band In Place (BIP) time.
- Decreased incidence of RAO complications at discharge, or 24 hours, whichever occurs first
- Decreased incidence of other complications associated with TRA, such as hematoma, bleeding, and oozing.
- Elimination or reduction in the need for additional equipment, such as Doppler units, plethysmographs and pulse oximeters to assess hemostasis band efficacy
- Facilitate arterial site management to the more specialized catheterization lab staff/personnel that are better trained to recognize complications that occur during (BIP) band in place time.
- Decreasing the workload to the staff by virtue of shortened band in place times and improve procedural throughput.
- Facilitate greater patient comfort resulting from decrease band in place time and faster wound healing.

In our recent pilot study of 180 patients<sup>11</sup> comparing the TR band (TRB) with and without the Statseal (SS), successful TRB deflation occurred at 43  $\pm$  14 minutes with SS and 160  $\pm$  43 minutes without SS (p<0.001). Minor hematomas occurred in 9 (10.3%) of TRB patients and 16 (17.2%) of SS patients (p=0.20). Radial artery occlusion occurred in 2% of patients in the SS group (p=NS). Outpatients randomized to SS were discharged on average 51  $\pm$  83.5 minutes earlier than control.

Thus, the Statseal was demonstrated to facilitate a rapid deflation protocol with the TRB, resulting in an earlier discharge, without evidence of significantly increased complication of hematomas or radial artery occlusion. However, critiques of these results suggested that the protocol of different times for first complete TRB deflation attempt (40 minutes with SS and 180 minutes without) biased the outcome of the study, even though the times were based on current practice. In addition, there was concern that the study was not sufficiently large to detect a potential increased risk of the rapid deflation protocol with SS.

The present study is designed to address these concerns by having an identical time to first deflation of 60 minutes between the two groups, and have a larger sample size to detect any excess in the risk of hematoma or radial artery occlusion.

#### II. DESCRIPTION OF THE STUDY DEVICE:

Recently, a new compound – potassium ferrate, in combination with a hydrophilic polymer which is formed in to a disc when compressed - has been used in conjunction with hemostasis bands to shorten compression times. This product (trade name StatSeal Advanced) is an FDA approved product comprised of a topical hydrophilic polymer and potassium ferrate disc, [Photo 1] formed by compression of the compound.



Photo 1: StatSeal Advanced Disc

When in the direct contact with even a small amount of blood, the compound forms an occlusive seal through simultaneous iron-mediated agglomeration of blood solids/proteins and rapid dehydration of the blood. Seal formation is independent of the clotting cascade, facilitating sealing regardless of anticoagulation / antiplatelet status of the patient. Following cessation of pressure being applied to the site, the remnants of StatSeal form what resemble a 'scab', and remains in place for 24 hours, covered with a band-aid or Tegaderm patch.

#### INDICATION FOR USE

StatSeal Advanced is a commercially available product in the United States, and is indicated for use on patients in whom the radial artery has been used to gain vascular access for a cardiovascular procedure.

### **DEVICE STORAGE AND ACCOUNTABILITY**

StatSeal Advanced is provided in a sterile, foil pouch to protect it from humidity / moisture. As with most medical products, it should be stored in a cool, dry, secure environment. StatSeal Advance will be provided at no charge by the manufacturer for use in the study.

Damaged devices will be returned to the manufacturer (Biolife, LLC, Sarasota,FL). All unused devices may be retained by the site for continued use, if they so choose.

### III. STUDY OBJECTIVE(S)

The primary objectives of this study are to evaluate the performance of StatSeal Advanced used in conjunction with the TR Band (SS) as compared to the TR Band without SS (TRB) relative to:

- 1. the Time to Hemostasis (TTH)
- 2. the incidence of access site or forearm hematoma
- 3. peri-procedural radial artery occlusion (RAO) at discharge or 24 hours, whichever occurs first, and;

Time to Hemostasis (TTH) is defined as the time period required to achieve hemostasis, more specifically the time during which the TRB is applying compressive force to the access site. The time period that a TRB is left on the wrist while totally deflated is not considered as part of the TTH time.

Hematoma are defined according to the EASY scale. (EASY Classification I-V, ranging from <5cm [I], 5-10cm [II], >10cm to forearm [III], above elbow [IV] and causing ischemia [V]).

Radial Artery Occlusion is defined as the absence of flow to the hand based upon plethysmography – pulse oximetry (Pleth-Ox) performed using the reverse Barbeau test.

Unlike the pilot trial of this device, the present study will have an identical time to first deflation of 60 minutes between the two groups, and have a larger sample size to detect any excess risk of hematoma or radial artery occlusion. The study may also help demonstrate a relatively low rate of radial artery occlusion with a rapid deflation protocol, even at lower doses of unfractionated heparin than currently recommended.

#### IV. STUDY DESIGN AND METHODOLOGY

### **STUDY DESIGN**

This study is a physician initiated, prospective, observational, two arm, randomized study to be performed at experienced 'Radial First' centers. A minimum of 100 patients having undergone successful radial catheterization will be enrolled in the study, 400 in each arm. Enrollment with continue at each site on discretion of the investigators until at least 100 patients are enrolled, with each center contributing a minimum of 50 patients. Clinicians will perform the catheterization in accordance with local standard practice, with no minimum amount of anticoagulation required.

#### **STUDY METHODS**;

<u>Patient Selection Criteria</u> Study subjects will be identified in the catheterization laboratory holding area and asked to sign the informed consent prior to their catheterization procedure before the administration of sedative agents.

#### Inclusion Criteria:

Patient undergoing diagnostic angiography or PCI via the radial artery

Patients with a Barbeau test prior to the procedure showing pattern A,B,or C.

### **Exclusion Criteria:**

Candidates for this study will be excluded if any **one** of the following criteria is true.

- Use of a radial sheath larger than 6 Fr (a 7Fr-in-6 Glidesheath Slender ® is allowed).
- Use of a hemostasis method or device besides the TR Band.
- Patients undergoing catheterization from the femoral, brachial, ulnar, or distal radial (snuffbox) artery approach.
- Use of an anticoagulant other than unfractionated heparin or bivalirudin.
- Any use of glycoprotein inhibitors or cangrelor.
- Use of sheathless guides.
- Any anticipated need for continued anticoagulation post-catheterization, including extended bivalirudin infusion.
- Any active treatment with oral anticoagulants continued during course of procedure.
- Presence of arteriovenous dialysis fistula in the ipsilateral arm.
- Any physical deformity or trauma / injury of either wrist that would prevent proper placement or function of the hemostasis band.
- Raynaud's syndrome or known peripheral vascular disease of the forearm.
- Inability of the patient to personally consent for the study. (no surrogate consent)
- History or presence of Radial Artery Occlusion.
- Barbeau test showing Pattern D.
- Cardiogenic shock or any clinical instability as assessed by the physician performing the procedure.

#### Transradial Catheterization Procedure

Transradial Cardiac Catheterization will be performed according to local practice standards with use of a sheath diameter of up to 6 Fr. (A 7Fr-in-6 Glidesheath Slender®, with an outer diameter of 6Fr is defined as a 6F sheath and is allowed.)

Patients will have their activated clotting time measured prior to sheath removal and at least 5 minutes following the initial dose of anticoagulant. Additional activated clotting time measurements for PCI would be expected as part of routine practice but not recorded. Vasodilators (nitroglycerin, verapamil) will be administered in accordance with local practice.

#### Timing of Subject Enrollment

A subject will be consented into the study prior to the administration of sedation prior to the procedure, and randomized at the conclusion of a successful procedure (after all anticoagulation and antiplatelet medication decisions have been made), at which time placement of the assigned device will occur. Eligibility for the study will be assessed at this time and the subject will have to meet all of the inclusion criteria and none of the exclusion criteria.

Randomization will be performed by means of sealed envelopes in randomization blocks of 100. Each envelope will be labeled by patient number containing device designation. Device designation in the envelopes will be random in occurrence. When a patient is officially enrolled (after successful completion of a TRA procedure), the envelope corresponding to that patient number in the Study Patient log will be pulled, opened, and the assignment revealed.

Each of the sites will be allotted an initial block of 100 envelopes, with sets of additional blocks of 100 envelopes as needed. On the discretion of the site principal investigator and the lead principal investigator, enrollment may continue until each site enrolls 50 patients. The maximum enrollment at any one site shall not exceed 50% of the total study enrollment.

#### End of Study Status / Effect of Withdrawals:

A subject will have completed the study when one of the following events is documented:

- 1. The patient is successfully enrolled, treated with a TRB, and completes all required follow up tests.
- 2. A subject withdraws consent to participate. Patients who withdraw from the study will have their data included to the extent allowable by law. As all study related procedures are expected to be completed on the day of the procedure or day after, subject withdrawal is not considered likely.

### **Protocol:**

#### Informed Consent:

Subjects must have read the contents of the written informed consent document, had all questions regarding the study adequately answered by study staff, and signed and dated the document prior to any study related activities.

Control patients: Patients will have a TR band applied over the arteriotomy site and inflated with 15-18ml of air. After aspirating and clearing the contents of the sheath, the radial sheath will be removed. The TR band will be deflated until bleeding occurs, and 2 ml of air will be reintroduced to provide hemostasis. Patent hemostasis will be documented with plethysmography and oximetry as described below within 5 minutes after band application and removal, and within 30 min of discharge or after 24 hours. The TR band will be left inflated and in place for 60 minutes following the procedure for all patients (regardless of diagnostic or PCI procedure), after which full deflation attempts will commence.

Statseal Protocol: Patients will have a Statseal Advance RAD (SS) disc applied after withdrawing the radial sheath 2-4 cm. A Tegaderm dressing will be applied to secure the disc position. The TR band will be applied over the SS disc with the center of the balloon (the green dot) over the center of the SS disc. The TR band will be inflated with 8cc of air (which is typically occlusive pressure), and the sheath removed. No deflation will occur immediately. After 20 minutes of pressure, 3 cc of air will be removed from the TR band. After an additional 40 minutes (60 minutes after procedure), the TR band will be completely deflated.

### For both groups of patients:

Aside from the 3 cc partial deflation at 20 minutes in the SS group, all other TR band deflations should be attempts to completely deflate the device. Should there be evidence of bleeding during deflation (pulsatile blood flow, rebleeding, ooze, hematoma formation), the TR band is to be re-inflated only to the extent required to control bleeding, and radial artery patency checked with plethysmography. Subsequent attempts at full TR band deflation should occur regularly and no less often than every 15 minutes.

### Pleth-Ox testing of radial artery patency (Reverse Barbeau):

Following hemostasis, a pulse oximeter should be placed on tip of the ipsilateral thumb or index (2<sup>nd</sup>) finger and left there for successive observation of pulsatile waveforms. Compress both the ulnar and radial arteries proximal or distal to the TR band to confirm sufficient pressure is present to close the artery. Release of pressure to the radial artery while maintaining ulnar compression will result in a normal distal waveform, diminished waveform, or absent waveform.

Absence of plethysmographic waveform is indicative of interruption of radial artery flow from radial artery occlusion. Investigators are recommended but not mandated to confirm diagnosed RAO with ultrasound if available.

#### Test methodology:

All Pleth-ox testing will be done by qualified personnel with results classified according to Barbeau test pattern classifications (for preprocedure assessment) or simplified classification (Normal, Diminished, or Absent waveform) (postprocedure assessments).

At the start of the TRA procedure, prior to radial artery cannulation, a baseline Pleth-ox exam will be performed for all patients and recorded on the CRF. Ulnar compression will be applied to confirm that the radial artery is patent. Patients with a type D pattern exam will be excluded from the study.

Following placement of the TRB system, reverse Pleth-Ox exams will be performed at the following time points with results recorded in the CRFs as the radial artery antegrade waveform being "normal", "diminished", or "absent".

- Within 5 minutes after initial TRB placement
- In the SS (StatSeal Advanced) group only, within 5 minutes after the first partial deflation (20 minutes after initial placement).
- At 60 minutes, following first full deflation attempt
- Within 5 minutes after successful full deflation of the TRB
- Within 30' of discharge or 24 hours post procedure (± 1 hour), whichever occurs first.

#### TR Band left in place (optional):

Following hemostasis, the completed deflated TR band may be left in place on the wrist for a period of time (<30 minutes) determined by local practice. This serves to remind the patient not to bend at the wrist and provides for the ability to rapidly reinflate the TR band should bleeding be detected. The TR band should be completed deflated in all cases. The duration the TR band is left in place should not be allowed to vary according to randomization assignment – each site investigator is asked to prespecify their protocol and apply the same time of deflated TR band to both groups.

[rest of page intentionally blank]



### V. STUDY DEFINITIONS AND OUTCOMES

### <u>Definitions of Baseline and Procedural Variables:</u>

Smoking: Active smoking or >20 pack year tobacco history.

Diabetes: Hgb A1C >6.5% or active medical treatment for diabetes.

Hypercholesterolemia: LDL >130 or on treatment with antilipemic agents.

Hypertension: >140/80 or on medical treatment for hypertension.

Diagnostic procedure: Involving diagnostic catheters only.

Interventional procedure: Involving an interventional wire and therapeutic ACT typically >50, including for fractional flow reserve measurement where a stent is not placed.

Single wall puncture: Use of micropuncture wire and anterior wall puncture only.

Double wall puncture: Use of double wall puncture and sheath withdrawal technique.

Puncture attempts: Number of forward advances of the needle (not puncture sites) needed to achieve access

Procedure Start Time: Time when lidocaine is administered, prior to first puncture attempt.

Procedure End Time: Time when sheath is removed.

### **Primary Efficacy Outcome:**

 Total Time to Hemostasis (TTH), defined as the total time the TR Band applies compressive force until successful hemostasis is achieved without complication. This is also described as the time of TR band inflation.

#### Secondary Efficacy Outcome:

 Time to discharge, defined as the time from the procedure completion to discharge of the patient

### Primary Safety Outcome:

Hematoma formation (EASY Classification I-V, ranging from <5cm [I], 5-10cm [II],</li>
 >10cm to forearm [III], above elbow [IV] and causing ischemia [V]).

#### Secondary Safety outcomes:

Radial artery occlusion, as detected by reverse Barbeau/Pleth-ox testing

#### VI. STUDY STATISTICAL PLAN:

This is a physician initiated, prospective, randomized, two-arm study, to be conducted at experienced 'Radial First' centers with the principal investigator having a (minimum) ten case experience using StatSeal Advanced. The primary analysis will be by intention-to-treat methodology.

The sample size of 100 patients is sufficient to have >95% power to detect an average expected difference of 20 minutes in time (60 min vs 80 min) to deflation of the TR band between the SS and TRB groups, using a two-sided alpha of 0.05, based on the results of the prior pilot study. The sample size is sufficient to have >95% power to detect an average expected difference of 20 minutes in time to discharge (170 min vs 190 min) between the SS and TRB groups, using a two-sided alpha of 0.05, based on the results of the prior pilot study adjusted for changes in protocol.

For safety outcomes, the sample size of 100 patients is estimated to have >95% power for noninferiority in radial artery occlusion rates, if the rates are consistent with what was seen in our prior pilot study (0% control vs 2% Statseal) at an absolute noninferiority margin of 0.5% and a two-sided alpha of 0.05. The study size will have >80% power for noninferiority in hematoma rates if the rates are consistent with what was seen in our prior pilot study (10% control vs 13% Statseal) at an absolute noninferiority margin of 3% and a two-sided alpha of 0.05.

Descriptive summary statistics will be presented for all study variables. Continuous variables will be displayed as means with standard deviations and medians with 75<sup>th</sup> and 25<sup>th</sup> percentiles. Categorical variables will be summarized as frequencies with their respective percentages with two-sided 95% exact confidence intervals of the percentages. Statistical comparisons for continuous variables will be performed using the Student's t test or Mann-Whitney U test, as appropriate. Comparisons for categorical variables will be performed using the Chi square test or Fisher exact test, as appropriate. A two-sided P value of 0.05 will be considered statistically significant.

Planned subgroup analyses will include analysis of the outcomes according to the following procedural characteristics:

- 1) Diagnostic vs PCI
- 2) Dose of heparin (<5000 units, >5000 units)

Multivariate analysis for hematoma formation and RAO are planned including but not limited to the factors of compression time, SS use, sheath size, heparin dose, closing ACT. An interim analysis will be performed when half of planned enrollment has been completed to review for futility or efficacy.

#### VII. ADVERSE EVENTS:

Reports of all adverse events will be made and recorded for the duration of the study, and categorized as specific to those complications associated with radial access, such as

hematoma, bleeding, RAO, and other vascular access complications. Those complications not related to vascular access will be stored locally only.

Adverse events will be recorded on CRFs and adjudicated by the site Principal Investigator as to their severity and whether or not directly, indirectly, or not connected to the study devices, and forwarded to the Data Center for entry in to the database.

#### Adverse Event

Any clinically relevant event that occurs during the performance of the study that puts the subject at additional risk of injury, whether foreseen or not, and requires additional care beyond that expected as a result of the study.

#### Adverse Device Event

An adverse event related to the use of the device. This includes adverse events resulting from insufficient or inadequate instructions for use, deployment, or operation, or any malfunction of the device. This definition also includes any event resulting from user error or from intentional misuse of the device by the investigator.

### Serious Adverse Event

A serious adverse event (SAE) is defined as an adverse event that:

- Led to death,
- Led to a serious deterioration in health that either,
  - o Resulted in a life-threatening illness or injury, or
  - o Resulted in a permanent impairment of a body structure or a body function, or
  - o Required in-patient hospitalization, or
  - Resulted in medical or surgical intervention to prevent life threatening illness or injury or permanent impairment to a body structure or a body function.

Note: This includes device deficiencies that might have led to a serious adverse event if (a) suitable action had not been taken or (b) intervention had not been made or (c) if circumstances had been less fortunate.

#### VIII. DATA MANAGEMENT

#### **Data Collection Process**

Data will be collected in an anonymized (coded) fashion using case report forms for each subject. CRFs will be transmitted to the data center for entry in to the database. Data may be collected by clinical research personnel assigned to the study, under the supervision of the investigator.

### Data Confidentiality

Subject data will be collected in an anonymous form. Each site will keep a confidential, site – only log of enrolled patients connecting their identity to a coded subject identifier. Each subject will be entered on the log along with procedure date and will be assigned a patient study number comprised of the site number and sequential subject number enrolled. This coded number will be used in the CRFs. For example, John Q Doe, the 12<sup>th</sup> patient enrolled at site

number 2, will be assigned study identifier 002-012. All activities will be performed in compliance with HIPPAA and Good Clinical Practice standards

#### Data Center

CRFs or coded anonymized data will be forwarded to the Data Center at the Long Beach VA Medical Center, checked for completeness, and entered in the Database as received. Incomplete forms will be returned to the study site for completion. Electronic submission of Data may be employed, but is not required.

See the "Study Statistical Plan" for a description of the plan.

### IX. ETHICAL, REGULATORY & ADMINISTRATIVE REQUIREMENTS

The devices being studied in this clinical plan, and the tests performed under it, are approved for marketing by the US-FDA for use as described and have been in use for TRA procedures at the participating institutions. FDA approval of the study is not required. No part of the study uses any device or test that is considered investigational.

#### Investigational Review Board Approvals.

Data from this study may be used for publication in the scientific literature, and therefor IRB approval is required. No patient may be enrolled until IRB approval is granted, and an Informed Consent approved by the IRB is signed by the subject.

#### Protocol Adherence and Amendments

Investigators will be required to adhere to the protocol requirements. Deviations or violations of the protocol may result in dismissal from the study.

#### Informed Consent

Each subject in the study must sign the informed consent agreeing to participation.

#### Alternatives to Participation

As a voluntary randomized study, the patient's alternative to participation is primarily to the local standard of care, typically involving the TR band, used per local protocol (typically 1-3 hours of application). SS devices may be used outside of the study depending on local practice and availability.

#### Enrollment in other studies

Simultaneous or dual enrollment in other investigative or observational protocols that do not involve vascular access, anticoagulation, or antiplatelet agents is expressly permitted. The interventions in this trial are not expected to significantly impact upon the outcomes of other protocols, however, the site investigator is responsible for ensuring that there is no conflict with dual enrollment from the standpoint of the other trial.

#### Study Activities

The Investigator is required to perform the study in accordance with the protocol and to use devices per their instructions for use.

### Follow-Up

There is no requirement for the subjects taking part in the study to be seen or examined for any follow up relative to the study following completion of activities described herein.

#### **CRFs**

CRFs will be completed for each subject. See Appendix 1 for the CRFs.

#### Records and Retention

Copies of all records will be retained by the investigator at each site for 2 years.

### (Model) Patient Informed Consent

See Appendix 2 for a model of the informed consent.

### Communication with the Principal Investigator:

All communication regarding the study should be routed directly to the Principal Investigator. Copies of all correspondence regarding the study should be maintained in the Site Investigator study file.

### Declaration of Helsinki & HIPPAA

The Principal Investigator will ensure that this study is performed in conformity with the Declaration of Helsinki, HIPPAA, and all local and national regulations.

### **Investigator Responsibilities**

- Adhere to all of the required elements of the Clinical Protocol
- Resolve queries in a timely manner
- · Participate in Investigator meetings and emails, if scheduled
- Comply with the Declaration of Helsinki
- Obtain written Informed Consent from each study participant before any study specific procedures are performed
- Complete all required case report forms (CRFs) for each subject
- Comply with all applicable regulations and codes of approvals from the site IRB and other Regulatory Authorities
- Notify the Principal Investigator of personnel changes that may affect the study protocol
- Retain all records and study files as required, after which the files may be destroyed.
- Allow direct access to source data/documents, including patient records, in case of monitoring, auditing and/or inspection by the IRB and/or other regulatory authority bodies.

### X. RISK BENEFIT ANALYSIS

### **General Risks and Presumed Benefits:**

Application of a hemostatic device in a setting absent an actual radial arteriotomy presents negligible risk to the subject. The only foreseen risk would be leaving an inflated band in place for an extended period of time. This risk is negligible provided the protocol is followed. An action of this nature would be considered a protocol violation.

Patients assigned to the SS group may enjoy less discomfort from the shorter length of time that the TRB is in place, presuming that the SS does reduce TRB compression time. Patient in the

TRB group may experience more attention to the arteriotomy wound and distal perfusion compared with those having been treated with a traditional protocol prior to the study.

Both groups having a planned first deflation time (60 minutes) that is earlier than the traditional 90-120 minute compression time of the TRB may be at an increased risk of hematoma formation. However, this risk should be minimized by the close attention to the vascular access site by the recovery room team. In addition, there is no standard deflation time specified in the TRB instructions for use, and prior studies have not detected a signal of harm with a 60 minute deflation time.

The potential benefit of subject participation is gratification from making a contribution to science helping to demonstrate the effectiveness of a new clinical method to achieve hemostasis following a radial artery procedure. This new method could potentially provide a safer, more efficient, and more effective hemostatic device for clinicians to use in treating patients undergoing the radial approach for cardiovascular procedures.

#### Risks related to Hemostasis Bands:

Currently marketed hemostasis bands have been associated with complications such as, but not limited to, skin irritation, radial artery occlusion, hematoma, pseudoaneurysm, failure to achieve hemostasis, and general wrist discomfort.

#### Risks Specific to the Study Device:

There are no known risks specific to the study device.

### Risk Mitigation:

Every effort will be made to mitigate risks in this Study. Those efforts include requiring investigators to be highly experienced Radialists, practicing at Radial First centers, and have used the study device in a minimum of ten cases.

Clinical monitoring will occur in real time to ensure the accurate collection and reporting of data, and ensure that the Site is in compliance with the clinical protocol requirements that mitigate risk such as patient entry criteria, use of the study device in accordance with instructions, and compliance with study test procedures and methods.

#### XI. REFERENCES:

- 1. Roffi M, Patrono C, Collet; ESC Scientific Document Group . 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315.
- 2. Cooper CJ, El-Shiekh RA, Cohen DJ, Blaesing L, Burket MW, Basu A, Moore JA. Effect of transradial access on quality of life and cost of cardiac catheterization: A randomized comparison. *Am Heart J*. 1999;138:430-436
- 3. Jolly SS, Amlani S, Hamon M, Yusuf S, Mehta SR. Radial versus femoral access for coronary angiography or intervention and the impact on major bleeding and ischemic events: a systematic review and meta-analysis of randomized trials. *Am Heart J*. 509;157:132-140

- 4. Safley DM, Amin AP, House JA, Baklanov D, Mills R, Giersiefen H, Bremer A, Marso SP. Comparison of costs between transradial and transfemoral percutaneous coronary intervention: a cohort analysis from the Premier research database. *Am Heart J*. 2013;165:303-309 e302
- Feldman DN, Swaminathan RV, Kaltenbach LA, Baklanov DV, Kim LK, Wong SC, Minutello RM, Messenger JC, Moussa I, Garratt KN, Piana RN, Hillegass WB, Cohen MG, Gilchrist IC, Rao SV. Adoption of radial access and comparison of outcomes to femoral access in percutaneous coronary intervention: an updated report from the national cardiovascular data registry (507-2012). Circulation. 2013;127:2295-2306
- 6. Bertrand OF, Rao SV, Pancholy S, Jolly SS, Rodes-Cabau J, Larose E, Costerousse O, Hamon M, Mann T. Transradial approach for coronary angiography and interventions: results of the first international transradial practice survey. *JACC Cardiovasc Interv*. 2010;3:1022-1031
- 7. Pancholy SB, Patel TM. Effect of duration of hemostatic compression on radial artery occlusion after transradial access. *Catheter Cardiovasc Interv.* 2012;79:78-81
- 8. Rao SV. Observations from a transradial registry: our remedies oft in ourselves do lie. *JACC Cardiovasc Interv*. 2012;5:44-46
- 9. Barbeau GR, Arsenault F, Dugas L, Simard S, Lariviere MM. Evaluation of the ulnopalmar arterial arches with pulse oximetry and plethysmography: comparison with the Allen's test in 1010 patients. *Am Heart J*. 504;147:489-493
- 10. Wang DS, Chu LF, Olson SE, Miller FJ, Valji K, Wong WH, Rose SC, Austin M, Kuo MD. Comparative Evaluation of Noninvasive Compression Adjuncts for Hemostasis in Percutaneous Arterial, Venous, and Arteriovenous Dialysis Procedures, Access Procedures. *Journal of Vascular and Interventional Radiology*. January 508; 19: 72-79.
- 11. Seto AH, Rollefson W, Patel MP, et al. Radial haemostasis is facilitated with a potassium ferrate haemostatic patch: the Statseal with TR Band assessment trial (STAT) EuroIntervention. 2018 Dec 7;14(11):e1236-e1242.

# **APPENDICES:**

Appendix 1: Sample Informed Consent

Appendix 2: CRF's